CLINICAL TRIAL: NCT04065204
Title: Metabolomic Analysis of Body Fluid of Medulloblastoma in Children Based on New Mass Spectrometry and Its Application in Clinical Diagnosis and Recurrence Monitoring
Brief Title: Metabolomic Analysis of Body Fluid of Medulloblastoma in Children
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Xinhua Hospital, Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Sponsor
Other Study IDs: XH-19-006
Record Dates: First submitted 2019-07-29; First posted 2019-08-22 (Actual); Last update posted 2019-09-23 (Actual); Status verified 2019-07

CONDITIONS: Pediatric Medulloblastoma
Keywords: Pediatric Medulloblastoma; Metabolomics; Radiation Therapy
MeSH Terms: conditions — Medulloblastoma

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Biospecimen Retention: Samples Without DNA — blood and urine
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Based on a new mass spectrometry system, body fluid samples were analyzed to verify the role of metabolite analysis in the diagnosis of pediatric medulloblastoma.

DETAILED DESCRIPTION:
Screening specific molecular metabolic markers for medulloblastoma after radiotherapy can improve the prediction of clinical diagnosis and prognosis of patients.The purpose of this study is to validate the role of metabolite analysis in the diagnosis of pediatric medulloblastoma based on the analysis of body fluid samples by a new mass spectrometry system.Based on the metabolic markers found by screening, the pathogenic mechanism of metabolic pathway blockade was explained, and the scientific basis for later treatment was put forward.

ELIGIBILITY:
Inclusion Criteria:

* The samples are previous biological sample database data;
* Sample collection time was 2017.05-2019.05;
* The patient's age is over 3 years old;
* KPS score ≥50 at the first diagnosis;
* The patient was a medulloblastoma patient who had received surgical treatment and had not received radiotherapy or chemotherapy before.

Exclusion Criteria:

* Recurrent patients;
* Patients suffered from other malignant tumors during radiotherapy;
* The body fluid samples or related clinical data are not perfect;
* Storage failure of body fluid samples such as lipid dissolution and hemolysis occurred.

Min Age: 3 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Different body fluid samples (blood,urine)of patients in each group are estimated to be 100 cases.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2019-06-01 (Actual); Primary Completion 2022-06-01 (Estimated); Study Completion 2022-06-01 (Estimated)

PRIMARY OUTCOMES:
Metabolic marker(Uracil in Da) | Changes of expression profiles of specific metabolic markers before and after radiotherapy,up to 3 months.
  1. By comparing the expression of small molecule metabolites in body fluids between normal control group and patients with medulloblastoma before radiotherapy, to find specific markers. 2. To evaluate the expression of this metabolic marker in medulloblastoma patients before and after radiotherapy.
Metabolic marker(4-Hydroxyproline in Da) | Changes of expression profiles of specific metabolic markers before and after radiotherapy,up to 3 months.
  1. By comparing the expression of small molecule metabolites in body fluids between normal control group and patients with medulloblastoma before radiotherapy, to find specific markers. 2. To evaluate the expression of this metabolic marker in medulloblastoma patients before and after radiotherapy.
Metabolic marker(Creatine in Da) | Changes of expression profiles of specific metabolic markers before and after radiotherapy,up to 3 months.
  1. By comparing the expression of small molecule metabolites in body fluids between normal control group and patients with medulloblastoma before radiotherapy, to find specific markers. 2. To evaluate the expression of this metabolic marker in medulloblastoma patients before and after radiotherapy.
Metabolic marker(Glutamic acid in Da) | Changes of expression profiles of specific metabolic markers before and after radiotherapy,up to 3 months.
  1. By comparing the expression of small molecule metabolites in body fluids between normal control group and patients with medulloblastoma before radiotherapy, to find specific markers. 2. To evaluate the expression of this metabolic marker in medulloblastoma patients before and after radiotherapy.

CONTACTS AND LOCATIONS:
Overall Officials: Mawei D Jiang, MD, Principal Investigator — Xin Hua Hospital affiliated to Shanghai Jiaotong University School of Medicine
Locations (1):
- The Department of Radiation Oncology, Xin Hua Hospital Affiliated to Shanghai Jiao Tong University School of Medicine, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Yes